CLINICAL TRIAL: NCT07297160
Title: Chimeric Antigen Receptor Treatment Targeting Lymphoma, Myeloma and Solid Tumors That Express CD70 (SEventY) CALySSEY
Brief Title: CD70.CAR for CD70+ Lymphoma, Myeloma and Solid Tumors
Acronym: CALySSEY
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Bilal Omer, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-55493 CALySSEY
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma; Myeloma; Solid Tumors; Sarcoma; Kidney Cancer
Keywords: Lymphoma; Myeloma; Solid Tumors; T cell; CD70.CAR T-cells; Blood Cancer; Lymph Gland Cancer
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell; Sarcoma; Kidney Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A - Lymphoma and Solid Tumors (Experimental): CD70.CAR: Three dose levels, and a possible dose level -1 in case of unexpected toxicity at dose level 1, will be evaluated for patients with lymphoma and solid tumors. Each patient will receive one T cell infusion. Dose levels will be defined based on number of transduced T cells measured by flow cytometry.
  The first three patients treated on the study will be adults 18 years of age or older, which can be treated in each cohort.
  Interventions: Biological: Dose Level -1; Biological: Dose Level 1 (starting dose level); Biological: Dose Level 2; Biological: Dose Level 3
- Treatment Arm B - Myeloma (Experimental): CD70.CAR: Three dose levels, and a possible dose level -1 in case of unexpected toxicity at dose level 1, will be evaluated for patients with myeloma. Each patient will receive one T cell infusion. Dose levels will be defined based on number of transduced T cells measured by flow cytometry.
  The first three patients treated on the study will be adults 18 years of age or older, which can be treated in each cohort.
  Interventions: Biological: Dose Level -1; Biological: Dose Level 1 (starting dose level); Biological: Dose Level 2; Biological: Dose Level 3

INTERVENTIONS:
Biological: Dose Level -1 — Dose Level -1: 3 x 10^5 cells/kg
Biological: Dose Level 1 (starting dose level) — Dose Level 1 (starting dose level): 1 x 10^6 cells/kg
Biological: Dose Level 2 — Dose Level 2: 3 x 10^6 cells/kg
Biological: Dose Level 3 — Dose Level 3: 1 x 10^7 cells/kg

SUMMARY:
This study is for patients who have a type of cancer that expresses the protein CD70, which includes lymphoma (lymph gland cancer), myeloma and solid tumors including some sarcomas and kidney cancers, and the cancer has come back or has not gone away after standard of care treatment.

As there are limited or no remaining standard treatments available to treat this cancer, patients are being asked to volunteer to be in a gene transfer research study using special immune cells to create a specialized immune cell that will recognize a protein called CD70 that is expressed on the outside surface of the tumor cells in the body.

This research study combines different ways of fighting disease by using T cells and "arming" them to recognize a specific protein on cancer cells. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells including tumor cells. T cells by themselves have been used to treat patients with cancers and have shown promise, but have not been strong enough to cure most patients.

The protein used in this study is called anti-CD70. It has been developed from human CD27 on normal T cells, since it is the natural binding partner that can connect with CD70. This anti-CD70 protein sticks to tumor cells when it binds to CD70. CD70 binders have been used to treat people with different types of cancers. For this study, anti-CD70 has been changed so that instead of floating free in the blood it is now joined to the T cells. When binder is joined to a T cell in this way it is called a chimeric receptor or "CAR T cell". The doctors then made another change to cause these T cells to kill any cell that has CD70. This causes the "CAR T cells" to kill blood cancer cells which are confirmed to have CD70.

In the laboratory, investigators have found that T cells work better if there are proteins added that stimulate T cells. The anti-CD70 (CD27) protein is unique because it can bind to CD70 on tumor cells but also stimulates the T cells that express it. Adding the CD27 makes the cells grow better and may help them to last longer in the body, thus giving the cells a better chance of killing the tumor cells.

These CD70 "CAR" T cells are investigational products not approved by the Food and Drug Administration.

The purpose of this study is to find a dose of CAR T cells that is safe, to learn what the side effects are and to see whether this therapy might help people with lymphoma (lymph gland cancer), myeloma and certain solid tumors including some sarcomas and kidney cancers.

DETAILED DESCRIPTION:
Blood will be collected from the patient to make CD70 CAR T cells. To make the T cells the blood will be stimulated with growth factors to make the T cells grow. To get the CD70 binder to attach to the surface of the T cell, investigators will insert the gene into the T cell. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps the investigators find the T cells in the blood after they are injected. To ensure the T cells grow well in the lab, investigators may add small amounts of medications that are often used to treat patients with cancer or other illnesses. These medications are washed off of the cells prior to injecting them into the patient's body. Because the patient will have received cells with a new gene in them, the patient will be followed for a total of 15 years to see if there are any long-term side effects of gene transfer. If the patient cannot visit the clinic, the patient may be contacted by the research coordinator or physician by phone or in other ways.

When the patient enrolls on this study, they will be assigned a dose of CD70 CAR T cells. Several studies suggest that the infused T cells need room to be able to proliferate (grow) and accomplish their functions and that this may not happen if there are too many other T cells in the blood. Because of that, the patient will receive two chemotherapy medications prior to receiving the CD70 CAR T cells. One medication is called cyclophosphamide and the other fludarabine. The patient will receive 3 daily doses of each drug, ending at least one day before receiving the CAR T cells. These drugs will decrease the numbers of the patients own T cells before infusion of the CD70 CAR T cells and also will help decrease the number of other cells that may interfere with the CAR T cells working well. Although there is no effect expected on the patient's tumor with the doses they will receive, these drugs are part of many regimens that are used to treat cancer. The investigators would prefer that the patient does not receive other chemotherapy or treatments for their cancer until 4 weeks after their cell infusion but the patient can do so if their doctor thinks it is medically necessary.

The patient will be given an injection of cells into the vein through an IV at the assigned dose. Before receiving the injection, the patient might be given a dose of Benadryl and Tylenol. The injection will take about 1-10 minutes. If no significant toxicities or signs of adverse/bad effects are seen right after infusion, the patient will be monitored for at least 2 hours post infusion. The patient will have to remain locally for at least 4 weeks after the infusion. If the patient experiences any side effects, they may have to be hospitalized for evaluation and management.

Medical Test Before Treatment:

* Physical exam and History
* Blood tests to measure blood cells, kidney and liver function
* Measurements of tumor by scans and/or bone marrow studies
* Testing of blood for certain viral infections
* An ultrasound of the heart to make sure the heart function is appropriate for the study if one has not been done recently

Medical Tests During and After Treatment:

* Physical exams and History
* Blood tests to measure blood cells, kidney and liver function
* Measurements of tumor by scans and/or bone marrow studies 4 weeks after the infusion

To learn more about the way the CD70 CAR T cells are working and how long they last in the body, extra blood will be drawn. The total amount on any day is about 10 teaspoons (50 mL) or no more than 3 mL per 2.2 pounds (3 ml per kilogram) body weight in children. This volume is considered safe but may be decreased if patient is anemic (decreased number of red blood cells). This blood may be drawn from a central line. Blood will be taken before starting chemotherapy a few days prior to the cell infusion. On the day patient receives the cells, blood will be taken before the cells are given and several hours afterwards. Other blood will be drawn one week after the infusion, 2 weeks, 3 weeks, 4 weeks 6 and 8 weeks after the infusion, at 3 months, at 6 months, at 9 months, at 1 year, every 6 months for 4 years, then yearly for a total of 15 years.

If the patient has a biopsy of their tumor or bone marrow studies in the future after completing this study, the investigators may ask to have a piece of tumor or bone marrow to look for CD70 CAR T cells.

In the event of the patient's death, the investigators will request permission to perform an autopsy to learn more about the effect of this experimental treatment on the tumor.

ELIGIBILITY:
PROCUREMENT INCLUSION CRITERIA:

• Diagnosis of relapsed/refractory T-cell acute lymphoblastic lymphoma (T-LLy), or T-non-Hodgkin Lymphoma (T-NHL, including Angioimmunoblastic T-cell lymphoma (AITL), Enteropathy-associated T-cell lymphoma (EATL), Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL), Peripheral T-cell lymphoma (PTCL) NOS, Anaplastic large cell lymphoma (ALCL), Adult T-cell lymphoma (lymphoma or chronic subtypes, Extranodal NK/T cell lymphoma, Mycosis fungoides (excluding Sezary Syndrome Stage IIB or higher) or multiply relapsed Hodgkin Lymphoma

OR

Patients with relapsed/refractory Renal Cell Carcinoma (RCC) OR sarcomas (for sarcoma only patients age 25 or younger are eligible)

OR

Patients with relapsed or refractory multiple myeloma (MM) that have failed or are ineligible for the 3 main classes of MM therapy ("triple class refractory")

(3 classes: 1. Immunomodulatory drugs, 2. proteosome inhibitors and 3. Anti-CD38 monoclonal antibodies).

* CD70 positive tumor with at least 26% CD70+ tumor cells by immunohistochemistry (staining can be pending at time of procurement)
* Age ≤75 years (except for sarcoma: only patients age ≤25 are eligible) NOTE: The first three (3) patients treated on the study will be adults (≥18 years of age)
* Hemoglobin ≥ 7.0 g/dL (can be transfused)
* If apheresis required to collect blood, PT and aPTT <1.5x ULN; Serum Creatinine < 2 x ULN; AST < 5 x ULN.

PROCUREMENT EXCLUSION CRITERIA:

* Active infection (bacterial, fungal or viral) requiring ongoing treatment without improvement.
* Known active infection with HIV or HTLV (collected blood will be sent for HIV/HTLV testing, separate testing prior to procurement not required). Patients with HIV are eligible if viral load is undetectable on therapy and CD4 count is >350 mm3.
* Active second cancer (except non-melanoma skin cancer or in situ breast cancer or cervical cancer) or other cancer treated ≤ 2 years prior to enrollment
* Ongoing treatment with immune suppression for prophylaxis/treatment of GVHD including high dose steroids (e.g., prednisone > 0.5 mg/kg/day).

TREATMENT INCLUSION CRITERIA:

• Diagnosis of relapsed/refractory T-cell acute lymphoblastic lymphoma (T-LLy), or T-non-Hodgkin Lymphoma (T-NHL, including Angioimmunoblastic T-cell lymphoma (AITL), Enteropathy-associated T-cell lymphoma (EATL), Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL), Peripheral T-cell lymphoma (PTCL) NOS, Anaplastic large cell lymphoma (ALCL), Adult T-cell lymphoma (lymphoma or chronic subtypes), , Extranodal NK/T cell lymphoma, Mycosis fungoides (excluding Sezary Syndrome Stage IIB or higher) or multiply relapsed Hodgkin Lymphoma

OR

Patients with relapsed/refractory Renal Cell Carcinoma (RCC) or sarcomas (for sarcoma only patients age 25 or younger are eligible)

OR

Patients with relapsed or refractory multiple myeloma (MM) that have failed or are ineligible for the 3 main classes of MM therapy ("triple class refractory") and also failed or ineligible for anti-BCMA therapies.

(3 classes: 1. Immunomodulatory drugs, 2. proteosome inhibitors and 3. Anti-CD38 monoclonal antibodies).

* CD70 positive tumor with at least 26% CD70+ tumor cells by immunohistochemistry (tissue)
* No systemic chemotherapy at least 2 weeks prior to treatment on study and must be recovered from all acute toxic effects of prior chemotherapy at time of treatment
* Age ≤75 years. (except for sarcoma: only patients age ≤25 are eligible) NOTE: The first three (3) patients treated on the study will be adults (≥18 years of age).
* Hemoglobin ≥ 7.0 g/dL (can be transfused)
* Total bilirubin < 3 times the upper limit of normal
* AST/ALT < 5 times the upper limit of normal
* Creatinine < 2 times the upper limit of normal
* Pulse oximetry of > 90% on room air
* Karnofsky or Lansky score of ≥60%
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. Male partner should use a condom.
* Informed Consent Obtained.

TREATMENT EXCLUSION CRITERIA:

* Received investigational anti-cancer agents < 28 days or 5 half-lives, whichever is shorter
* Received any tumor vaccines within the previous 6 weeks
* Pregnant or lactating
* Uncontrolled infection with HIV, or HTLV. Patients with HIV are eligible if viral load is undetectable on therapy and CD4 count is >350 mm3.
* Clinically significant bacterial, fungal, or viral infection requiring ongoing therapy without improvement.
* Cardiac abnormalities: Cardiac echocardiography with LVEF<50%; Cardiac dysfunction NYHA III or IV; Clinically significant pericardial effusion. Confirmation of absence of these conditions must be obtained within 6 months of treatment.
* Use of serotherapy with Campath or Anti-Thymocyte Globulin (ATG) within the last 28 days
* Use of Donor Lymphocyte Infusion (DLI) or other cellular therapy product within 28 days.
* Acute GVHD ≥ Grade 2 or moderate to severe (formerly extensive) chronic GVHD.
* High dose steroids >1 mg/kg within the preceding 5 days or currently receiving >0.5 mg/kg/day prednisone equivalent.
* Bulky CNS or mediastinal disease that significantly increases potential risks (e.g. airway obstruction, TIAN) in the estimation of a principal investigator.

Ages: 0 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2044-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) rate | 4 weeks post infusion
  Toxicity for all patients will be evaluated using the NCI Common Toxicity Criteria Scale with the exception of CRS and immune effector cell associated neurotoxicity (ICANS). CRS and ICANS will be graded per ASTCT consensus grading criteria.

SECONDARY OUTCOMES:
Overall response rate | 6-8 weeks post infusion
  The study will use the revised response criteria for malignant lymphoma to evaluate response in patients with T-cell lymphoma and the international myeloma working group response assessment guidelines for MM. Patients with solid tumors (RCC and sarcomas) will be assessed by iRECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Omer, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas